CLINICAL TRIAL: NCT00855868
Title: Evaluation of the Ability of a Novel [18F] Amyloid Ligand ([18F]-AV-45) to Distinguish Patients With a Clinical Diagnosis of Alzheimer's Disease From Cognitively Normal Elderly Individuals
Brief Title: Ability Of ([18F]-AV-45) PET Scan to Distinguish Alzheimer's Disease Subjects From Cognitively Normal Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Collaborators: American College of Radiology Imaging Network (Network); General Electric (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ACRIN PA 4003
Record Dates: First submitted 2009-03-02; First posted 2009-03-05 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-06

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid imaging; Positron Emission Tomography; 18F-AV-45; florbetapir F 18; Diagnostic imaging
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir; 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: florbetapir F 18 — 370 MBq (10 mCi), intravenous (IV) injection, single dose
  Other Names: 18F-AV-45; Amyvid; florbetapir
Drug: [11C]-PIB — 555 MBq (15 mCi), IV injection, single dose [11C]-PIB
  Other Names: C-11 PIB

SUMMARY:
This study will evaluate the performance characteristics of a novel [18F] amyloid detection ligand (18F]-AV-45) with respect to its ability to distinguish patients with clinically-diagnosed probable Alzheimer's disease from cognitively normal elderly subjects and to independently compare its diagnostic performance characteristics with the ability of [11C]PIB to correctly categorize the same subjects.

SPECIFIC HYPOTHESES

1. Individuals with a clinical diagnosis of probable Alzheimer's disease will have increased brain retention of [18F]-AV-45 compared to cognitively normal elderly individuals.
2. There will be no clinically meaningful difference in the amyloid retention performance characteristics of [18F]-AV-45 and [l1C]PIB.

DETAILED DESCRIPTION:
15 patients with a clinical diagnosis of probable Alzheimer's disease and 15 cognitively normal elderly control subjects will receive both [18F]-AV-45 and [11C]PIB to compare the diagnostic performance characteristics of each amyloid ligand to distinguish AD from normal subjects. In addition to clinical diagnostic category, ligand retention will be evaluated with respect to measures of symptom severity and cerebrospinal fluid levels of amyloid and tau.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects: mini-mental state examination (MMSE) 27-30, clinical dementia rating (CDR) = 0, no symptoms of depression
* Alzheimer's subjects: MMSE 18-26, CDR >=0.5, University of Pennsylvania Alzheimer's Disease Center consensus diagnosis of probable AD, absence of abnormalities on MRI

Exclusion Criteria:

* other neurological disease
* evidence of MRI abnormality
* psychiatric disorder
* alcohol abuse
* clinically significant lab abnormalities
* residence in nursing facility
* participation in clinical trial with experimental medication in past 1 month

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Alzheimer's Disease: Mini-mental state examination (MMSE) 18-26, clinical dementia rating (CDR) >=0.5, University of Pennsylvania Alzheimer's Disease Center consensus diagnosis of probable AD, absence of abnormalities on MRI and age 55-90
- Healthy Controls: Cognitively normal with MMSE of 27 or higher, CDR=0, no symptoms of depression and age 55-90 years.
Period: Overall Study
Arm/Group | Alzheimer's Disease | Healthy Controls
Started | 13 | 15
Completed | 12 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alzheimer's Disease | Healthy Controls | Total
Number analyzed (Participants) | 13 | 15 | 28
Age Continuous [Mean (Standard Deviation); unit: years] | 69.8 (9.88) | 71.5 (9.23) | 70.7 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Differences in Standard Uptake Value Ratio (SUVR) for Frontal Cortex/Cerebellum and Whole Brain/Cerebellum of the Positron Emission Tomography (PET) Scan With [18F]-AV-45 for Probable Alzheimer's Disease (AD) Versus Cognitively Normal Subjects.
Description: Standardized Uptake Value ratio (SUVR) as measured in this study indicates the ratio of tracer uptake in the frontal cortex relative to the cerebellum or the ratio of tracer uptake in the whole brain relative to the cerebellum.
Time Frame: 28 d
Measure: Mean (Standard Deviation); unit: SUVR
Arm/Group | Alzheimer's Disease | Healthy Controls
Number analyzed (Participants) | 12 | 14
SUVR
  Frontal cortex to cerebellum SUVR | 1.33 (.20) | 1.00 (.18)
  Whole brain to cerebellum SUVR | 1.38 (.15) | 1.06 (.17)

ADVERSE EVENTS:
Arm/Group | Alzheimer's Disease | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 4/13 | 1/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alzheimer's Disease (N=13) | Healthy Controls (N=15)
Visual Disturbance (Eye disorders) | 1 (1) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No